CLINICAL TRIAL: NCT03607656
Title: The Effect of Traditional Chinese Treatment Combined Adjuvant Chemotherapy in IIIb and IIIc Gastric Cancer: A Randomized Controlled Trial
Brief Title: The Effect of Traditional Chinese Treatment Combined Adjuvant Chemotherapy in IIIb and IIIc Gastric Cancer
Acronym: CHANGE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: RenJi Hospital (Other); Jiangsu Province Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, zhaoaiguang, Principal Investigator, Clinical Professor, Shanghai University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LONGHUA-2018-SH
Record Dates: First submitted 2018-07-01; First posted 2018-07-31 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Gastric Cancer Stage IIIB; Gastric Cancer Stage IIIC
MeSH Terms: conditions — Stomach Neoplasms | interventions — Oxaliplatin; Capecitabine; S 1 (combination); Docetaxel; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TCM combines CapOX/SOX/S-1+D/FLOT (Experimental): Traditional Chinese Medicine oral taken twice a day for at least 3 months combined with chemotherapy.
  The chemotherapy can choose intravenous oxaliplatin 130 mg/m(2) on day 1 plus oral capecitabine 1000 mg/m(2) twice daily on days 1-14, every 21 days; or intravenous oxaliplatin 100 mg/m(2) on day 1 plus oral S-1 40mg/m(2) twice daily on days 1-14, every 21 days; or intravenous docetaxel 40mg/m(2) on day 1 plus oral S-1 40mg/m(2) twice daily on days 1-14, every 21 days; or intravenous docetaxel 50mg/m(2) on day 1 plus intravenous oxaliplatin 85 mg/m(2) on day 1 plus 5-FU intravenously CIV24h on day 1, every 14 days; Each participant shoud take eight (8) cycles of chemotherapy.
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Other: TCM; Drug: S-1; Drug: Docetaxel; Drug: 5-FU
- CapOX/SOX/S-1+D/FLOT (Active Comparator): The chemotherapy can choose intravenous oxaliplatin 130 mg/m(2) on day 1 plus oral capecitabine 1000 mg/m(2) twice daily on days 1-14, every 21 days; or intravenous oxaliplatin 100 mg/m(2) on day 1 plus oral S-1 40mg/m(2) twice daily on days 1-14, every 21 days; or intravenous docetaxel 40mg/m(2) on day 1 plus oral S-1 40mg/m(2) twice daily on days 1-14, every 21 days; or intravenous docetaxel 50mg/m(2) on day 1 plus intravenous oxaliplatin 85 mg/m(2) on day 1 plus 5-FU intravenously CIV24h on day 1, every 14 days; Each participant shoud take eight (8) cycles of chemotherapy.
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Drug: S-1; Drug: Docetaxel; Drug: 5-FU

INTERVENTIONS:
Drug: Oxaliplatin — Oxaliplatin powder injection
Drug: Capecitabine — Capecitabine tablet
Other: TCM — TCM decoction orally taken twice a day for at least 3 months
  Arms: TCM combines CapOX/SOX/S-1+D/FLOT
Drug: S-1 — S-1 capsule
Drug: Docetaxel — Docetaxel injection
Drug: 5-FU — 5-FU injection

SUMMARY:
This is a randomized, open-label study done in 3 hospitals in China. Patients with stage IIIB and IIIC gastric cancer who undergo curative D2 gastrostomy will be randomly assigned after surgery to receive adjuvant chemotherapy with oxaliplatin and capecitabine, or adjuvant chemotherapy combined Traditional Chinese treatment. The primary outcome was disease-free survival and 3-year disease-free survival rate in the intention-to-treat population.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the Traditional Chinese Medicine combined adjuvant chemotherapy in the treatment of stage IIIb and IIIc gastric cancer through randomized controlled trial.

Metastasis and recurrence is the primary cause in decreasing the survival time of gastric cancer patients who experienced radical operation. Among whom, patients with stage IIIB and IIIC are especially in high risk of metastasis and recurrence, result in a significant poor survival time than patients with earlier stages.

Oxaliplatin with capecitabine is the standard adjuvant chemotherapy for curative D2 gastrostomy gastric cancer, contribute the 3-year disease free survival rate of 74% in ITT, and 61% in stage IIIB sub-group. Meanwhile, Traditional Chinese Medicine (TCM) treatment has been used for thousands of years in Chinese clinical practices. In China, the clinical curative effect of TCM in the treatment of gastric cancer has been part of affirmation. Some reports with large samples of clinical research show that the TCM is effective and safety for gastric cancer.In order to evaluate efficacy on TCM combined adjuvant chemotherapy in IIIB and IIIC gastric cancer, we design this randomized, open-label study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven gastric carcinoma with radical operation, TNM (primary tumor, regional nodes, metastasis) stage IIIb or IIIc （The Eighth Edition American Joint Committee on Cancer [AJCC] gastric cancer staging）;
* Karnofsky performance status higher than 70;
* Adequate hepatic, renal, cardio and hematologic function;
* With patients' consent and comply to long term follow-up.

Exclusion Criteria:

* Gastrectomy beyond D2, or TNM stage beyond Ⅲb and Ⅲc;
* Histological type beyond gastric carcinoma;
* Conversion chemotherapy before surgery;
* Concurrent cancer;
* Women of gravid or lactating; patients with mental illness;
* Uncontrolled significant comorbid conditions.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
3-year Disease Free Survival rate | 36 months
  The rate refers to cases that see first tumor metastasis or recurrence or death of any cause from randomization.

SECONDARY OUTCOMES:
Safety （adverse effects） | 36 months
  Using NCI-CTC standard to record adverse effects of chemotherapy and treatments.
EORTC QLQ-C30 scale | 36 months
  Using the EORTC QLQ-C30 scale (European Organization for Research on Treatment of Cancer Quality of Life Questionnaire-Core 30) to evaluate the quality of life of patients. The scale includes 14 aspects: physical functioning, role functioning, emotional functioning, cognitive functioning, social functioning, fatigue, nausea/vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial problem, with each aspect scores from one point to four points (lower points represent a better quality of life), and a general quality of life scores from one point to seven points (higher points represent a better quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: Aiguang Zhao, M.D.,Ph.D, Principal Investigator — Shanghai University of Traditional Chinese Medicine
Locations (1):
- Longhua Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bang YJ, Kim YW, Yang HK, Chung HC, Park YK, Lee KH, Lee KW, Kim YH, Noh SI, Cho JY, Mok YJ, Kim YH, Ji J, Yeh TS, Button P, Sirzen F, Noh SH; CLASSIC trial investigators. Adjuvant capecitabine and oxaliplatin for gastric cancer after D2 gastrectomy (CLASSIC): a phase 3 open-label, randomised controlled trial. Lancet. 2012 Jan 28;379(9813):315-21. doi: 10.1016/S0140-6736(11)61873-4. Epub 2012 Jan 7. PMID 22226517
- [Background] Xu Y, Zhao AG, Li ZY, Zhao G, Cai Y, Zhu XH, Cao ND, Yang JK, Zheng J, Gu Y, Han YY, Zhu YJ, Yang JZ, Gao F, Wang Q. Survival benefit of traditional Chinese herbal medicine (a herbal formula for invigorating spleen) for patients with advanced gastric cancer. Integr Cancer Ther. 2013 Sep;12(5):414-22. doi: 10.1177/1534735412450512. Epub 2012 Jul 9. PMID 22781545
- [Derived] Li Z, Zhang G, Cao N, Xu J, Dong J, Li J, Zhu X, Xu Y, Han C, Wang R, Xia X, Zhao G, Huan X, Fan J, Zhao A. Effects of traditional Chinese medicine collaborative model (TCMCM) combined with adjuvant chemotherapy on IIIb and IIIc gastric cancer: a protocol for a randomized controlled trial. Trials. 2022 Jan 21;23(1):68. doi: 10.1186/s13063-022-06013-5. PMID 35063002